CLINICAL TRIAL: NCT02892149
Title: Phase 3, Randomized, Open-Label, Active-Controlled Study Evaluating the Efficacy and Safety of Oral Vadadustat for the Maintenance Treatment of Anemia in Subjects With Dialysis-Dependent Chronic Kidney Disease (DD-CKD) (INNO2VATE-CONVERSION)
Brief Title: Efficacy and Safety Study to Evaluate Vadadustat for the Maintenance Treatment of Anemia in Participants With Dialysis-dependent Chronic Kidney Disease (DD-CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0017; 2016-001360-11 (EudraCT Number)
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Dialysis-Dependent Chronic Kidney Disease
Keywords: AKB-6548; Chronic kidney disease; anemia; CKD; chronic renal insufficiency; renal impairment; erythropoietin; kidney; renal; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; efficacy; safety; Phase 3; cardiovascular; DD-CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Masking Description: Sponsor was blinded during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vadadustat (Experimental)
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — Oral dose administered once daily for ≥36 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Darbepoetin alfa — Subcutaneous or intravenous dose administered for ≥36 weeks. Initial dose based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
A multicenter, randomized, open-label, active-controlled Phase 3 study for the maintenance treatment of anemia in participants with dialysis-dependent chronic kidney disease (DD-CKD)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled Phase 3 study of the efficacy and safety of Vadadustat versus Darbepoetin alfa for the maintenance treatment of anemia in participants with DD-CKD

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Receiving chronic maintenance dialysis (either peritoneal or hemodialysis) for end-stage kidney disease for at least 12 weeks prior to Screening
* Currently maintained on erythropoiesis-stimulating agent therapy, with a dose received within 6 weeks prior to or during Screening
* Mean Screening hemoglobin between 8.0 and 11.0 grams per deciliter (g/dL) (inclusive) in the US and between 9.0 and 12.0 g/dL (inclusive) outside of the US
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20% during Screening

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease or participants with active bleeding or recent blood loss
* Uncontrolled hypertension
* Red blood cell transfusion within 8 weeks prior to randomization
* Anticipated to recover adequate kidney function to no longer require dialysis
* Severe heart failure at Screening (New York Heart Association Class IV)
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure, or stroke within 12 weeks prior to or during Screening
* Hypersensitivity to Vadadustat, Darbepoetin alfa, or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3554 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (233):
- United States (109):
  - Research Site, Huntsville, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Pine Bluff, Arkansas
  - Research Site, Anaheim, California
  - Research Site #1, Bakersfield, California
  - Research Site #2, Bakersfield, California
  - Research Site, Canyon Country, California
  - Research Site, Chula Vista, California
  - Research Site, Downey, California
  - Research Site, El Centro, California
  - Research Site, Escondido, California
  - Research Site, Fairfield, California
  - Research Site, Glendale, California
  - Research Site #1, Granada Hills, California
  - Research Site #2, Granada Hills, California
  - Research Site, La Habra, California
  - Research Site, La Mesa, California
  - Research Site, Lakewood, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site #1, Montebello, California
  - Research Site, Monterey Park, California
  - Research Site, Newhall, California
  - Research Site #1, Northridge, California
  - Research Site #2, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site #1, San Dimas, California
  - Research Site #2, San Dimas, California
  - Research Site, Simi Valley, California
  - Research Site, Tarzana, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site #1, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - AMPM Research Clinic, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Augusta, Georgia
  - Research Site #1, Columbus, Georgia
  - Research Site #2, Columbus, Georgia
  - Research Site #1, Lawrenceville, Georgia
  - Research Site #2, Lawrenceville, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Statesboro, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Fort Wayne, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Monroe, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Takoma Park, Maryland
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Columbus, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Gallup, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, Astoria, New York
  - Research Site, Flushing, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Yonkers, New York
  - Research Site, Asheville, North Carolina
  - Research Site #1, Charlotte, North Carolina
  - Research Site #2, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site #1, New Bern, North Carolina
  - Research Site #2, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site #1, Chattanooga, Tennessee
  - Research Site #2, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Duncanville, Texas
  - Research Site, El Paso, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site #2, San Antonio, Texas
  - Research Site, St. George, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Hampton, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
- Argentina (8):
  - Research Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research Site, Junín, Buenos Aires
  - Research Site, Pergamino, Buenos Aires
  - Research Site, Sarandí, Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
  - Research Site, San Luis
- Australia (8):
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Launceston, Tasmania
  - Research Site, Box Hill, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Nedlands, Western Australia
- Brazil (17):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Feira de Santana, Estado de Bahia
  - Research Site, Itabuna, Estado de Bahia
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Maringá, Paraná
  - Research Site, Canoas, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Criciúma, Santa Catarina
  - Research Site, Joinville, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, São Bernardo do Campo, São Paulo
  - Research Site, São José do Rio Preto, São Paulo
  - Research Site, São Paulo, São Paulo
- Bulgaria (15):
  - Research Site, Byala
  - Research Site, Cherven Bryag
  - Research Site, Dobrich
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vidin
  - Research Site, Vratsa
- Canada (6):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- France (5):
  - Research Site, Marseille, Bouches-du-Rhône
  - Research Site, Bordeaux, Gironde
  - Research Site, Reims, Marne
  - Research Site, Saint-Priest-En-Jarez, Pays de la Loire Region
  - Research Site, Paris
- Germany (4):
  - Research Site, Villingen-Schwenningen, Baden-Wurttemberg
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Berlin
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rishon LeZiyyon
- Italy (6):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Siena
- Mexico (4):
  - Research Site, Pachuca, Hidalgo
  - Research Site, Zapopan, Jalisco
  - Research Site, Morelia, Michoacán
  - Research Site, Culiacán, Sinaloa
- Poland (5):
  - Research Site, Biała Podlaska
  - Research Site, Golub-Dobrzyń
  - Research Site, Kołobrzeg
  - Research Site, Lodz
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Beja
  - Research Site, Leiria
  - Research Site, Loures
- Russia (6):
  - Research Site #2, Kemerovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novorossiysk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Serbia (7):
  - Research Site #1, Belgrade
  - Research Site #2, Belgrade
  - Research Site #3, Belgrade
  - Research Site #4, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Zaječar
- South Korea (8):
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Seoul
- Ukraine (12):
  - Research Site, Brovary
  - Research Site #1, Cherkassy
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Mykolaiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr
- United Kingdom (5):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, London, Greater London
  - Research Site, Stevenage, Hertfordshire
  - Research Site, Kettering, Leicestershire
  - Research Site, Doncaster, South Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chertow GM, Eckardt KU, Sarnak MJ, Winkelmayer WC, Agarwal R, Minga T, Luo W, Burke SK. Safety and Efficacy of Vadadustat for the Treatment of CKD-Related Anemia within and outside the United States. J Am Soc Nephrol. 2025 Oct 1;36(10):1984-1997. doi: 10.1681/ASN.0000000708. Epub 2025 May 13. PMID 40359056
- [Derived] Sarnak MJ, Agarwal R, Boudville N, Chowdhury PCP, Eckardt KU, Gonzalez CR, Kooienga LA, Koury MJ, Ntoso KA, Luo W, Parfrey PS, Vargo DL, Winkelmayer WC, Zhang Z, Chertow GM. Vadadustat for treatment of anemia in patients with dialysis-dependent chronic kidney disease receiving peritoneal dialysis. Nephrol Dial Transplant. 2023 Sep 29;38(10):2358-2367. doi: 10.1093/ndt/gfad074. PMID 37096396
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Eckardt KU, Agarwal R, Aswad A, Awad A, Block GA, Bacci MR, Farag YMK, Fishbane S, Hubert H, Jardine A, Khawaja Z, Koury MJ, Maroni BJ, Matsushita K, McCullough PA, Lewis EF, Luo W, Parfrey PS, Pergola P, Sarnak MJ, Spinowitz B, Tumlin J, Vargo DL, Walters KA, Winkelmayer WC, Wittes J, Zwiech R, Chertow GM. Safety and Efficacy of Vadadustat for Anemia in Patients Undergoing Dialysis. N Engl J Med. 2021 Apr 29;384(17):1601-1612. doi: 10.1056/NEJMoa2025956. PMID 33913638

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4944 participants were screened for entry into the study. Of these, 3554 participants were enrolled and randomized in the study.
Groups:
- Vadadustat: Participants were randomized to receive Vadadustat at an initial oral dose of 300 milligrams per day (mg/day). Thereafter, Vadadustat was taken once daily on an outpatient basis. Up-and-down titration to 150, 300, 450, and 600 mg (available tablet strength was administered as the appropriate number of 150 mg tablets) was allowed during the study based on hemoglobin (Hb) level measurements to maintain target Hb levels.
- Darbepoetin Alfa: Participants were randomized to Darbepoetin alfa at an initial dose that was based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics (SmPC) for all other investigational sites (non-US) for adult participants with chronic kidney disease on dialysis. For participants already on Darbepoetin alfa, the initial dosing regimen in the study was based on the prior dosing regimen.
Period: Overall Study
Arm/Group | Vadadustat | Darbepoetin Alfa
Started | 1777 | 1777
Completed | 1425 | 1421
Not Completed | 352 | 356
Not completed — Death | 262 | 278
Not completed — Withdrawal by Subject | 53 | 47
Not completed — Lost to Follow-up | 37 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 1777 | 1777 | 3554
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (13.86) | 58.4 (13.84) | 58.1 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 787 | 773 | 1560
  Male | 990 | 1004 | 1994
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 30 | 49
  Asian | 76 | 99 | 175
  Black or African American | 432 | 444 | 876
  Native Hawaiian or Other Pacific Islander | 13 | 6 | 19
  White | 1135 | 1096 | 2231
  Not Reported | 52 | 52 | 104
  Reported as Other | 42 | 45 | 87
  Multiple | 8 | 5 | 13
Average hemoglobin [Mean (Standard Deviation); unit: Grams per deciliter (g/dL)] | 10.249 (0.8502) | 10.229 (0.8245) | 10.239 (0.8374)
Number of Participants on Different Types of Dialysis [Count of Participants; unit: Participants] — Dialysis assessment was performed at least 12 weeks prior to the first screening visit. A participant could be included for both peritoneal dialysis and hemodialysis at Baseline (i.e., not mutually exclusive parameters). Population: Participants initiating chronic dialysis was summarized in the Safety Population (INNO2VATE) which included all participants from the INNO2VATE population who received 1 or more doses of study drug.
  Participants
    Peritoneal Dialysis: number analyzed (Participants) | 1768 | 1769 | 3537
    Peritoneal Dialysis | 137 | 143 | 280
    Hemodialysis: number analyzed (Participants) | 1768 | 1769 | 3537
    Hemodialysis | 1652 | 1633 | 3285
Mean Years Since Chronic Dialysis Initiated [Mean (Standard Deviation); unit: Years] — Population: Participants with missing chronic dialysis initiation date were not included for the analysis.
  Years
    number analyzed (Participants) | 1775 | 1777 | 3552
    (all) | 4.004 (4.0224) | 3.941 (4.0144) | 3.973 (4.0180)
Number of Participants with History of Diabetes [Count of Participants; unit: Participants] | 794 | 820 | 1614
Number of Participants with NYHA Functional Classification of Heart Failure [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification serves as a fundamental descriptor of heart failure. NYHA heart failure classes are as follows: Class 0 (no congestive heart failure [CHF]), Class I (No symptoms and no limitation in ordinary physical activity), Class II (Mild symptoms and slight limitation during ordinary activity), Class III (Marked limitation in activity due to symptoms, even during less-than-ordinary activity), and Class IV (Severe limitations. Experiences symptoms even while at rest). NYHA class IV is also an exclusion criteria.
  Participants
    NYHA Class 0 | 1243 | 1221 | 2464
    NYHA Class I | 268 | 307 | 575
    NYHA Class II | 202 | 192 | 394
    NYHA Class III | 59 | 53 | 112
    NYHA Class IV | 0 | 0 | 0
    NYHA Class Missing | 5 | 4 | 9
Number of Participants with Any History of Heart Failure [Count of Participants; unit: Participants]
  Yes | 361 | 368 | 729
  No | 990 | 985 | 1975
  Missing | 426 | 424 | 850

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) to the Average Over the Primary Efficacy Period (Weeks 24 to 36)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Primary Efficacy Period was calculated as the average Hb value over Weeks 24 to 36. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with Baseline hemoglobin concentration (<10.0 versus ≥10.0 g/dL), geographic region (United States [US] versus European Union [EU] versus Rest of World [ROW]), and New York Heart Association congestive heart failure (NYHA CHF) class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 24 to 36
Population: Randomized Population: All participants randomized. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 1777 | 1777
Grams per deciliter (g/dL) | 0.19 (0.032) | 0.36 (0.032)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — Establishment of non-inferiority was based on a margin of -0.75 g/dL applied to the difference in mean change: Vadadustat minus Darbepoetin alfa; Least squares mean difference = -0.17, 95% CI 2-sided [-0.23 to -0.10], Standard Error of Mean 0.03

2. Primary Outcome: Median Time to First Major Adverse Cardiovascular Event (MACE)
Description: MACE was defined as all-cause mortality, non-fatal myocardial infarction (MI), or non-fatal stroke. The primary safety outcome was positively adjudicated first MACE, which was defined as any death, Endpoint Adjudication Committee (EAC)-confirmed non-fatal MI, or EAC-confirmed non-fatal stroke occurring between the first dose date and each participant's last participation date. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0017 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 170 weeks
Population: Safety Population (INNO2VATE): All participants from the INNO2VATE population who received 1 or more doses of study drug. Only those participants with MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 333 | 353
Weeks | 48.86 [26.43 to 79.71] | 48.00 [22.43 to 75.57]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0017 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per Food and Drug Administration [FDA]) and 1.30 (per European Medicines Agency [EMA]); p = 0.4745, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.828 to 1.117]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 355 and 377 respectively; median time to first event (Q1, Q3) = 46.14 (24.71, 77.14) weeks versus 47.00 (22.43, 74.43) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4877, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.833 to 1.113]

3. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Efficacy Period (Weeks 40 to 52)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Secondary Efficacy Period was calculated as the average Hb value over Weeks 40 to 52. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with Baseline hemoglobin concentration (<10.0 versus ≥10.0 g/dL), geographic region (US versus EU versus ROW), and NYHA CHF class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 40 to 52
Population: Randomized Population. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 1777 | 1777
g/dL | 0.23 (0.035) | 0.41 (0.033)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Least squares mean difference = -0.18, 95% CI 2-sided [-0.25 to -0.12], Standard Error of Mean 0.04

4. Secondary Outcome: Median Time to First MACE Plus Hospitalization for Heart Failure or Thromboembolic Event Excluding Vascular Access Thrombosis
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Hospitalization for EAC adjudicated heart failure included presentation of participants to an acute care facility requiring an overnight hospitalization (change in calendar day) with an exacerbation of heart failure requiring treatment. EAC confirmed thromboembolic events for this secondary outcome measure included arterial thrombosis, deep vein thrombosis, and pulmonary embolism. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0017 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 170 weeks
Population: Safety Population (INNO2VATE). Only those participants with MACE plus hospitalization for heart failure or thromboembolic event excluding vascular access thrombosis were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 391 | 418
Weeks | 43.29 [21.86 to 73.14] | 45.21 [22.29 to 73.86]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0017 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.3718, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.832 to 1.097]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first MACE plus hospitalization for heart failure or thromboembolic event Excluding vascular access thrombosis for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 420 and 449 respectively; median time to first event (Q1, Q3) = 42.07 (21.50, 71.14) weeks versus 45.29 (22.29, 72.43) weeks, respectively; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4096, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.840 to 1.096]

5. Secondary Outcome: Median Time to First Cardiovascular MACE
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Cardiovascular MACE analysis differed from the primary MACE endpoint as it included only deaths adjudicated by the EAC as cardiovascular deaths (i.e, only EAC-confirmed cardiovascular deaths) in addition to first events of non-fatal MI or non-fatal stroke. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0017 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 170 weeks
Population: Safety Population (INNO2VATE). Only those participants with cardiovascular MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 209 | 228
Weeks | 44.57 [23.29 to 81.86] | 43.57 [20.71 to 73.93]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0017 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.3875, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.777 to 1.131]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first cardiovascular MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 225 and 242 respectively; median time to first event (Q1, Q3) = 43.29 (21.71, 77.14) weeks versus 45.79 (21.14, 73.86) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.5007, Gray's test; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.795 to 1.144]

6. Secondary Outcome: Median Time to First Cardiovascular Death
Description: Cardiovascular death included EAC adjudicated fatal MI, pump failure, sudden death, presumed sudden death, fatal stroke, fatal pulmonary embolism, cardiovascular procedure-related death, other cardiovascular death, and presumed cardiovascular death. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0017 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 170 weeks
Population: Safety Population (INNO2VATE). Only those participants with cardiovascular death were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 141 | 150
Weeks | 46.14 [29.43 to 79.00] | 47.64 [24.57 to 74.14]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0017 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.6281, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.761 to 1.203]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first cardiovascular death for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 150 and 160 respectively; median time to first event (Q1, Q3) = 43.71 (27.43, 77.14) weeks versus 49.29 (24.43, 74.07) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.6284, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.766 to 1.195]

7. Secondary Outcome: Median Time to First All-cause Mortality
Description: Only events that were positively adjudicated and confirmed by the EAC were included in the MACE analyses. INNOVATE MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Results and statistical analysis from study AKB-6548-CI-0017 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0016 and AKB-6548-CI-0017 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to 170 weeks
Population: Safety Population (INNO2VATE). Only those participants with all-cause mortality were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 276 | 290
Weeks | 50.79 [30.29 to 80.50] | 50.43 [26.14 to 78.86]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0017 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.5811, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.816 to 1.136]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0016 (NCT02865850) and AKB-6548-CI-0017 (NCT02892149). Time to first all-cause mortality for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 291 and 310 respectively; median time to first event (Q1, Q3) = 50.00 (29.71, 79.00) weeks versus 49.57 (25.86, 77.29) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.30 (per EMA); p = 0.4878, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.812 to 1.118]

8. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Proportion of Participants With an Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory - Time to Achieve Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory - Mean Change in Hb Between Baseline (Mean Pretreatment Hb) and the Primary Evaluation Period (Mean Hb From Weeks 24 to 36) Stratified by Pre-baseline Erythropoiesis-stimulating Agent (ESA) Exposure
Time Frame: Baseline; Weeks 24 to 36
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory - Mean Monthly Dose of Intravenous (IV) Elemental Iron Administered in Participants Who Have Received IV Iron
Time Frame: Up to Week 52
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving IV Iron Therapy
Time Frame: Up to Week 52
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving Red Blood Cells (RBCs) Transfusion(s)
Time Frame: Up to Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 170 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported in study AKB-6548-CI-0017 (NCT02892149). Of the participants randomized, 3537 participants were included in the Safety population (1768 and 1769 participants in the Vadadustat and Darbepoetin alfa treatment groups, respectively). 17 randomized participants did not receive treatment.
Arm/Group | Vadadustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 276/1768 | 290/1769
Serious Adverse Events (participants affected / at risk) | 973/1768 | 1032/1769
Other Adverse Events (participants affected / at risk) | 964/1768 | 993/1769
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=1768) | Darbepoetin Alfa (N=1769)
Pneumonia (Infections and infestations) | 140 | 119
Fluid overload (Metabolism and nutrition disorders) | 98 | 98
Sepsis (Infections and infestations) | 76 | 88
Acute myocardial infarction (Cardiac disorders) | 81 | 78
Hyperkalaemia (Metabolism and nutrition disorders) | 55 | 76
Cardiac arrest (Cardiac disorders) | 49 | 60
Cardiac failure congestive (Cardiac disorders) | 45 | 50
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 56 | 38
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 44 | 50
Septic shock (Infections and infestations) | 44 | 45
Atrial fibrillation (Cardiac disorders) | 44 | 37
Cellulitis (Infections and infestations) | 43 | 38
Anaemia (Blood and lymphatic system disorders) | 35 | 37
Osteomyelitis (Infections and infestations) | 31 | 39
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 27 | 42
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 34 | 29
Coronary artery disease (Cardiac disorders) | 28 | 32
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 26 | 33
Hypotension (Vascular disorders) | 29 | 30
Non-cardiac chest pain (General disorders) | 34 | 22
Cardio-respiratory arrest (Cardiac disorders) | 28 | 26
Peritonitis (Infections and infestations) | 21 | 32
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 | 26
Device related infection (Infections and infestations) | 25 | 23
Gangrene (Infections and infestations) | 24 | 23
Urinary tract infection (Infections and infestations) | 15 | 32
Metabolic encephalopathy (Nervous system disorders) | 20 | 25
Cardiac failure acute (Cardiac disorders) | 18 | 26
Hypertensive urgency (Vascular disorders) | 19 | 25
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 22 | 20
Hypertension (Vascular disorders) | 20 | 22
Blood loss anaemia (Blood and lymphatic system disorders) | 16 | 24
Hypoglycaemia (Metabolism and nutrition disorders) | 22 | 18
Syncope (Nervous system disorders) | 22 | 18
Death (General disorders) | 24 | 14
Acute left ventricular failure (Cardiac disorders) | 13 | 23
Influenza (Infections and infestations) | 20 | 15
Fall (Injury, poisoning and procedural complications) | 17 | 18
Staphylococcal sepsis (Infections and infestations) | 16 | 18
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 16 | 18
Mental status changes (Psychiatric disorders) | 11 | 23
Hypertensive emergency (Vascular disorders) | 16 | 18
Staphylococcal bacteraemia (Infections and infestations) | 17 | 15
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Bronchitis (Infections and infestations) | 12 | 19
Cerebrovascular accident (Nervous system disorders) | 14 | 16
Chest pain (General disorders) | 14 | 15
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Encephalopathy (Nervous system disorders) | 13 | 12
Ischaemic stroke (Nervous system disorders) | 13 | 12
Hypertensive crisis (Vascular disorders) | 12 | 13
Cardiogenic shock (Cardiac disorders) | 10 | 14
End stage renal disease (Renal and urinary disorders) | 15 | 9
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 11 | 12
Deep vein thrombosis (Vascular disorders) | 13 | 10
Peripheral vascular disorder (Vascular disorders) | 13 | 10
Myocardial infarction (Cardiac disorders) | 10 | 12
Arteriovenous graft site infection (Infections and infestations) | 8 | 14
Gastroenteritis (Infections and infestations) | 8 | 14
Femur fracture (Injury, poisoning and procedural complications) | 15 | 7
Angina unstable (Cardiac disorders) | 8 | 13
Cardiac failure (Cardiac disorders) | 9 | 11
Abdominal pain (Gastrointestinal disorders) | 8 | 12
Bacteraemia (Infections and infestations) | 9 | 11
Endocarditis (Infections and infestations) | 5 | 15
Vascular access malfunction (Injury, poisoning and procedural complications) | 10 | 10
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 7 | 13
Seizure (Nervous system disorders) | 6 | 14
Transient ischaemic attack (Nervous system disorders) | 15 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Angina pectoris (Cardiac disorders) | 8 | 11
Arteriovenous fistula site infection (Infections and infestations) | 12 | 7
Clostridium difficile colitis (Infections and infestations) | 7 | 12
Diverticulitis (Infections and infestations) | 9 | 10
Pneumonia bacterial (Infections and infestations) | 7 | 12
Diabetic foot (Skin and subcutaneous tissue disorders) | 7 | 12
Pancreatitis acute (Gastrointestinal disorders) | 10 | 8
Postoperative wound infection (Infections and infestations) | 5 | 13
Colitis (Gastrointestinal disorders) | 8 | 9
Gastritis (Gastrointestinal disorders) | 9 | 8
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 12
Hip fracture (Injury, poisoning and procedural complications) | 6 | 11
Ventricular tachycardia (Cardiac disorders) | 9 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 9
Cholelithiasis (Hepatobiliary disorders) | 7 | 9
Atrial flutter (Cardiac disorders) | 6 | 9
Bradycardia (Cardiac disorders) | 4 | 11
Cholecystitis acute (Hepatobiliary disorders) | 6 | 9
Hepatic enzyme increased (Investigations) | 7 | 8
Azotaemia (Renal and urinary disorders) | 10 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 8
Pericardial effusion (Cardiac disorders) | 2 | 12
Device related sepsis (Infections and infestations) | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Extremity necrosis (Vascular disorders) | 8 | 6
Cardiopulmonary failure (Cardiac disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Abscess limb (Infections and infestations) | 7 | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 6 | 7
Alanine aminotransferase increased (Investigations) | 7 | 6
Peripheral ischaemia (Vascular disorders) | 7 | 6
Ascites (Gastrointestinal disorders) | 3 | 9
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 7
Asthenia (General disorders) | 6 | 6
Sudden death (General disorders) | 3 | 9
Aspartate aminotransferase increased (Investigations) | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Left ventricular failure (Cardiac disorders) | 4 | 7
Impaired gastric emptying (Gastrointestinal disorders) | 6 | 5
Intestinal ischaemia (Gastrointestinal disorders) | 8 | 3
Pancreatitis (Gastrointestinal disorders) | 5 | 6
Pyrexia (General disorders) | 3 | 8
Diabetic foot infection (Infections and infestations) | 3 | 8
Transaminases increased (Investigations) | 8 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 7
Haematoma (Vascular disorders) | 9 | 2
Shock haemorrhagic (Vascular disorders) | 8 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 8
Mitral valve incompetence (Cardiac disorders) | 2 | 8
Colitis ischaemic (Gastrointestinal disorders) | 5 | 5
Cholecystitis (Hepatobiliary disorders) | 7 | 3
Catheter site infection (Infections and infestations) | 4 | 6
Localised infection (Infections and infestations) | 5 | 5
Wound infection (Infections and infestations) | 5 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 7
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 5
Haemorrhagic stroke (Nervous system disorders) | 3 | 7
Device dislocation (Product Issues) | 6 | 4
Aortic stenosis (Vascular disorders) | 3 | 7
Jugular vein thrombosis (Vascular disorders) | 3 | 7
Shock (Vascular disorders) | 5 | 5
Intestinal obstruction (Gastrointestinal disorders) | 7 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 7
Appendicitis (Infections and infestations) | 4 | 5
Staphylococcal infection (Infections and infestations) | 4 | 5
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 4 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Hepatic encephalopathy (Nervous system disorders) | 3 | 6
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 5 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Nephrogenic anaemia (Blood and lymphatic system disorders) | 6 | 2
Myocardial ischaemia (Cardiac disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 6 | 2
Duodenal ulcer (Gastrointestinal disorders) | 6 | 2
Catheter site thrombosis (General disorders) | 5 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 4 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 4 | 4
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 | 4
Dizziness (Nervous system disorders) | 4 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 | 4
Pulseless electrical activity (Cardiac disorders) | 4 | 3
Ventricular fibrillation (Cardiac disorders) | 3 | 4
Inguinal hernia (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 2 | 5
Impaired healing (General disorders) | 6 | 1
Systemic inflammatory response syndrome (General disorders) | 4 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 6
Cytomegalovirus infection (Infections and infestations) | 3 | 4
Osteomyelitis acute (Infections and infestations) | 1 | 6
Peritonitis bacterial (Infections and infestations) | 3 | 4
Urosepsis (Infections and infestations) | 1 | 6
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 6
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4
Cerebral haemorrhage (Nervous system disorders) | 3 | 4
Cerebral infarction (Nervous system disorders) | 3 | 4
Presyncope (Nervous system disorders) | 2 | 5
Acute kidney injury (Renal and urinary disorders) | 4 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dry gangrene (Vascular disorders) | 3 | 4
Peripheral artery thrombosis (Vascular disorders) | 4 | 3
Pancytopenia (Blood and lymphatic system disorders) | 4 | 2
Arrhythmia (Cardiac disorders) | 1 | 5
Atrioventricular block complete (Cardiac disorders) | 2 | 4
Chronic left ventricular failure (Cardiac disorders) | 3 | 3
Supraventricular tachycardia (Cardiac disorders) | 2 | 4
Tachycardia (Cardiac disorders) | 1 | 5
Chronic gastritis (Gastrointestinal disorders) | 2 | 4
Gastritis erosive (Gastrointestinal disorders) | 4 | 2
Ileus (Gastrointestinal disorders) | 4 | 2
Melaena (Gastrointestinal disorders) | 4 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3
Arthritis bacterial (Infections and infestations) | 2 | 4
Fungal peritonitis (Infections and infestations) | 3 | 3
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Graft thrombosis (Injury, poisoning and procedural complications) | 5 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 4
Perirenal haematoma (Injury, poisoning and procedural complications) | 3 | 3
Pubis fracture (Injury, poisoning and procedural complications) | 3 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 3
Liver function test increased (Investigations) | 2 | 4
Carotid artery stenosis (Nervous system disorders) | 1 | 5
Haemorrhage intracranial (Nervous system disorders) | 5 | 1
Hypertensive encephalopathy (Nervous system disorders) | 3 | 3
Device malfunction (Product Issues) | 4 | 2
Haematuria (Renal and urinary disorders) | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cardiac failure chronic (Cardiac disorders) | 5 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 4
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 3
Sinus node dysfunction (Cardiac disorders) | 2 | 3
Hyperparathyroidism (Endocrine disorders) | 3 | 2
Hyperparathyroidism secondary (Endocrine disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 | 2
Catheter site haemorrhage (General disorders) | 2 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 4
Gastroenteritis viral (Infections and infestations) | 3 | 2
Infected skin ulcer (Infections and infestations) | 3 | 2
Pyelonephritis (Infections and infestations) | 2 | 3
Streptococcal bacteraemia (Infections and infestations) | 2 | 3
Subcutaneous abscess (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 4
Head injury (Injury, poisoning and procedural complications) | 3 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Rib fracture (Injury, poisoning and procedural complications) | 2 | 3
Vascular graft complication (Injury, poisoning and procedural complications) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Brain injury (Nervous system disorders) | 4 | 1
Uraemic encephalopathy (Nervous system disorders) | 3 | 2
Chronic kidney disease (Renal and urinary disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Arteriosclerosis (Vascular disorders) | 2 | 3
Hypovolaemic shock (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 4
Peripheral artery occlusion (Vascular disorders) | 1 | 4
Steal syndrome (Vascular disorders) | 4 | 1
Coronary artery occlusion (Cardiac disorders) | 2 | 2
Pericarditis (Cardiac disorders) | 1 | 3
Tricuspid valve incompetence (Cardiac disorders) | 3 | 1
Cataract (Eye disorders) | 3 | 1
Diverticular perforation (Gastrointestinal disorders) | 3 | 1
Faecaloma (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 3 | 1
Generalised oedema (General disorders) | 3 | 1
Sudden cardiac death (General disorders) | 3 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 2 | 2
Bronchitis viral (Infections and infestations) | 3 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 3
Gas gangrene (Infections and infestations) | 0 | 4
Intervertebral discitis (Infections and infestations) | 2 | 2
Large intestine infection (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Pneumonia viral (Infections and infestations) | 2 | 2
Pseudomonal bacteraemia (Infections and infestations) | 2 | 2
Vascular access site infection (Infections and infestations) | 0 | 4
Viral infection (Infections and infestations) | 3 | 1
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 | 4
Delayed graft function (Injury, poisoning and procedural complications) | 1 | 3
Eschar (Injury, poisoning and procedural complications) | 1 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 4
Troponin increased (Investigations) | 2 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 3
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Status epilepticus (Nervous system disorders) | 2 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 1 | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 3
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 3
Hospitalisation (Surgical and medical procedures) | 1 | 3
Malignant hypertension (Vascular disorders) | 2 | 2
Splenic infarction (Blood and lymphatic system disorders) | 1 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 3 | 0
Enteritis (Gastrointestinal disorders) | 3 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 3 | 0
Peptic ulcer (Gastrointestinal disorders) | 3 | 0
Physical deconditioning (General disorders) | 2 | 1
Treatment noncompliance (General disorders) | 2 | 1
Liver injury (Hepatobiliary disorders) | 1 | 2
Abdominal abscess (Infections and infestations) | 1 | 2
Acute hepatitis B (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 2 | 1
Candida infection (Infections and infestations) | 1 | 2
Cholecystitis infective (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 3
Diabetic gangrene (Infections and infestations) | 0 | 3
Endocarditis bacterial (Infections and infestations) | 2 | 1
Endocarditis staphylococcal (Infections and infestations) | 1 | 2
Escherichia bacteraemia (Infections and infestations) | 3 | 0
Infection (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 2 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 1 | 2
Staphylococcal abscess (Infections and infestations) | 2 | 1
Tooth abscess (Infections and infestations) | 2 | 1
Tracheobronchitis (Infections and infestations) | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 2 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Postoperative hypotension (Injury, poisoning and procedural complications) | 2 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 2
Shunt thrombosis (Injury, poisoning and procedural complications) | 2 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 2
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 3
Calciphylaxis (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Altered state of consciousness (Nervous system disorders) | 3 | 0
Brain hypoxia (Nervous system disorders) | 1 | 2
Brain oedema (Nervous system disorders) | 1 | 2
Cerebellar infarction (Nervous system disorders) | 2 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 2
Embolic stroke (Nervous system disorders) | 1 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 2
Hypoglycaemic encephalopathy (Nervous system disorders) | 2 | 1
Lacunar infarction (Nervous system disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Renal cyst (Renal and urinary disorders) | 2 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Brachiocephalic vein occlusion (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 2 | 1
Superior vena cava syndrome (Vascular disorders) | 2 | 1
Venous stenosis (Vascular disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 2
Atrial tachycardia (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 2
Coronary artery thrombosis (Cardiac disorders) | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 2 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 2 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 2 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Catheter site pain (General disorders) | 1 | 1
Complication associated with device (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 1 | 1
Surgical failure (General disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 1
Arthritis infective (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 2
Breast abscess (Infections and infestations) | 0 | 2
Catheter site abscess (Infections and infestations) | 1 | 1
Cellulitis staphylococcal (Infections and infestations) | 2 | 0
Chronic hepatitis B (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 2
Escherichia pyelonephritis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 1
Graft infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 2
Klebsiella infection (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 2 | 0
Perineal abscess (Infections and infestations) | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 1
Pneumonia serratia (Infections and infestations) | 1 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Renal graft infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Scrotal abscess (Infections and infestations) | 2 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 1
Vascular device infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Vulval abscess (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 1
Renal lymphocele (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 2
Vascular access site complication (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 1
False positive investigation result (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Coma (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 2
Myoclonus (Nervous system disorders) | 0 | 2
Neurotoxicity (Nervous system disorders) | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 1
Device occlusion (Product Issues) | 1 | 1
Thrombosis in device (Product Issues) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 2
Penile vascular disorder (Reproductive system and breast disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Therapy cessation (Surgical and medical procedures) | 1 | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 2
Superior vena cava occlusion (Vascular disorders) | 0 | 2
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic artery perforation (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 0 | 1
Intracardiac mass (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve calcification (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Pericarditis uraemic (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery thrombosis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal wall oedema (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diabetic gastropathy (Gastrointestinal disorders) | 0 | 1
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Uraemic gastropathy (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Cardiac death (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Hernia pain (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Necrosis (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Soft tissue inflammation (General disorders) | 1 | 0
Strangulated hernia (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Ulcer (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Contrast media reaction (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Renal transplant failure (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Achromobacter infection (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Atypical mycobacterial pneumonia (Infections and infestations) | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Bullous impetigo (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Cerebral septic infarct (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cystitis klebsiella (Infections and infestations) | 1 | 0
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Emphysematous cholecystitis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Fournier's gangrene (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Giardiasis (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 1 | 0
Implant site cellulitis (Infections and infestations) | 1 | 0
Incision site abscess (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Mycobacterium fortuitum infection (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis bacterial (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paraspinal abscess (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Perinephric abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pseudomonas peritonitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyuria (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Rhodococcus infection (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 0 | 1
Septic encephalopathy (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Splenic infection (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Systemic infection (Infections and infestations) | 0 | 1
Testicular abscess (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis viral (Infections and infestations) | 0 | 1
Transplant abscess (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Vessel puncture site infection (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 0 | 1
Viral sepsis (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Dialysis disequilibrium syndrome (Injury, poisoning and procedural complications) | 0 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 | 1
Incision site swelling (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 | 0
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural shock (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site rupture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Ammonia increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Influenza B virus test positive (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone metabolism disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Hungry bone syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Amputation stump pain (Nervous system disorders) | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Central nervous system lupus (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebral artery thrombosis (Nervous system disorders) | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hyperammonaemic encephalopathy (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Jugular vein occlusion (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Microvascular cranial nerve palsy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Post cardiac arrest syndrome (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device extrusion (Product Issues) | 1 | 0
Device failure (Product Issues) | 0 | 1
Device leakage (Product Issues) | 1 | 0
Device physical property issue (Product Issues) | 0 | 1
Patient-device incompatibility (Product Issues) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary bladder rupture (Renal and urinary disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Testicular oedema (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Living in residential institution (Social circumstances) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Haemodialysis (Surgical and medical procedures) | 0 | 1
Large intestinal polypectomy (Surgical and medical procedures) | 1 | 0
Procoagulant therapy (Surgical and medical procedures) | 1 | 0
Vascular access placement (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Brachiocephalic vein stenosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Distributive shock (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0
Neurogenic shock (Vascular disorders) | 0 | 1
Obstructive shock (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Subclavian vein occlusion (Vascular disorders) | 0 | 1
Subclavian vein stenosis (Vascular disorders) | 0 | 1
Subgaleal haemorrhage (Vascular disorders) | 1 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Vascular stenosis (Vascular disorders) | 1 | 0
Vasculitis necrotising (Vascular disorders) | 0 | 1
Vein rupture (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=1768) | Darbepoetin Alfa (N=1769)
Hypertension (Vascular disorders) | 175 | 232
Diarrhoea (Gastrointestinal disorders) | 226 | 173
Headache (Nervous system disorders) | 160 | 134
Fall (Injury, poisoning and procedural complications) | 136 | 144
Nausea (Gastrointestinal disorders) | 148 | 131
Hyperkalaemia (Metabolism and nutrition disorders) | 123 | 137
Hypotension (Vascular disorders) | 124 | 119
Vomiting (Gastrointestinal disorders) | 119 | 123
Dialysis related complication (Injury, poisoning and procedural complications) | 99 | 122
Cough (Respiratory, thoracic and mediastinal disorders) | 99 | 120
Upper respiratory tract infection (Infections and infestations) | 98 | 108
Pain in extremity (Musculoskeletal and connective tissue disorders) | 84 | 113
Urinary tract infection (Infections and infestations) | 100 | 93
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 79 | 111
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 80 | 107
Nasopharyngitis (Infections and infestations) | 92 | 84
Back pain (Musculoskeletal and connective tissue disorders) | 71 | 92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT02892149/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02892149/SAP_001.pdf